CLINICAL TRIAL: NCT05586633
Title: The Efficacy of Ultrasound-guided Deep Paravertebral-periforaminal Ozone Injection in the Treatment of Patients With Chronic Low Back Pain
Brief Title: The Efficacy of Ultrasound-guided Ozone Injection in the Treatment of Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Sefa Gümrük Aslan, Principal Investigator, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32
Record Dates: First submitted 2022-08-14; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Low Back Pain, Posterior Compartment
Keywords: Low Back Pain; periforaminal ozon injection; transforaminal steroid injection; ultrasound guided injection
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep paravertebral- periforaminal ozone injection (Active Comparator)
  Interventions: Procedure: deep paravertebral periforaminal ozone injeciton
- transforaminal steroid injeciton (Active Comparator)
  Interventions: Procedure: transforaminal steroid injeciton

INTERVENTIONS:
Procedure: deep paravertebral periforaminal ozone injeciton — Deep paravertebral periforaminal ozone injection was administered to the patients in the ozone injection group 4 times under ultrasound guidance, 10 ug/ml 5ml twice a week in the first week and 15 ug/ml 5ml twice a week in the second week.
  Patients will be evaluated according to the study criteria at the beginning, at 15 days, 1 month, and 2 months. Physical examination findings were evaluated before starting the treatment and at the 2nd month follow-up.
  Arms: deep paravertebral- periforaminal ozone injection
Procedure: transforaminal steroid injeciton — Transforaminal epidural steroid injection group, steroid (dexamethasone 8mg/2ml 2ml) injection was performed under the guidance of fluoroscopy.
  Patients will be evaluated according to the study criteria at the beginning, at 15 days, 1 month, and 2 months. Physical examination findings were evaluated before starting the treatment and at the 2nd month follow-up.
  Arms: transforaminal steroid injeciton

SUMMARY:
Low back pain is a common disorder that every individual in the society is likely to meet throughout his/her life. Low back pain lasting longer than 12 weeks is defined as chronic low back pain and causes serious disability in the community. Conservative, pharmacological, interventional and surgical treatment options are available in its treatment. In this study, it was aimed to determine the effects of ultrasound-guided deep paravertebral periforaminal ozone injection treatment on physical examination, functional independence, quality of life and pain scores in patients with chronic low back and leg pain and to compare it with transforaminal epidural steroid injection treatment.

DETAILED DESCRIPTION:
A total of 50 patients were included in the study. Deep paravertebral periforaminal ozone injection was administered to the patients in the ozone injection group 4 times under ultrasound guidance, 10 ug/ml 5ml twice a week in the first week and 15 ug/ml 5ml twice a week in the second week. In the transforaminal epidural steroid injection group, steroid (dexamethasone 8mg/2ml 2ml) injection was performed under the guidance of fluoroscopy. The patients in both groups were offered a home exercise program for therapeutic waist and abdominal muscles to do during the treatment follow-up period. Patients' quality of life was evaluated with SF-36(Short Form-36), pain scores with VAS(Visüel Analog Scala) and functional evaluations with ODI(Oswestry Disability Index) at 15 days, 1 month, and 2 months. Physical examination findings were evaluated before starting the treatment and at the 2nd month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Back and leg pain lasting longer than 3 months
* Diagnosis of lumbar disc herniation with advanced imaging techniques after anamnesis, - physical examination and laboratory examinations
* Continuation of complaints despite conservative treatment before
* Regular participation in the study voluntarily

Exclusion Criteria:

* Being pregnant and breastfeeding
* History of lomber surgery
* Peripheral neuropathy (diabetes, alcoholism...)
* Cauda equina syndrome or progressive neurologic deficit in the lower extremity
* Neurogenic bladder/bowel syndrome
* Arterial vascular disease-Vascular claudication
* Spinal stenosis, spondylolysis, spondylolisthesis
* Local infection at the injection site
* Presence of bleeding diathesis
* Neuro-degenerative diseases
* Uncontrolled diabetes, hypertension
* History of malignancy
* Uncontrolled psychiatric illness
* BMI over 40
* Allergy to injection substances

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
PAİN-Visual Analog Scala (VAS) | 2nd week, 4th week, 8th week pain change
  Visual Analog Scala (VAS), patients are asked to circle the number between 0 and 10 that fits best to their pain intensity. Severity of pain was assessed VAS using the standard 10 cm (back pain and leg pain) with 0 meant "no pain" at one end, and 10 meant "unbearable pain" at the other end.
Quality of life - Short Form-36 (SF-36) | 2nd week, 4th week, 8th week quality of life change
  Satisfaction assessed by the SF-36. Short Form (SF-36) was used to investigate the quality of life of the patients.The reliability and validity of the Turkish version of SF-36 has been demonstrated. SF-36 consists of 36 questions on eight different subscales including physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, energy and fatigue, vitality, social functioning, role limitations due to emotional problems and general mental health. Each subscale of SF-36 is scored between 0 and 100, and higher scores show better Quality of life.
Oswestry Disability Index (ODI) | 2nd week, 4th week, 8th week pain change
  In the ODI questionnaire, the effect of low back pain on activities of daily living is questioned. In the test, which consists of 10 questions in total, the patient's pain intensity, the effects of pain on personal care, walking, lifting weights, standing, sitting, sleeping, sexual life, social life and traveling are questioned. The patient can get a minimum of 0 and a maximum of 5 points from each question. The maximum score to be taken from the test is 50. The patient's score is found by dividing the total score of the patient by 50, which is the maximum score, and calculating the percentage. (Patient's score ÷ maximum score × 100). Accordingly, it is calculated how much the patient's life activities are affected.
Physical examination-Lumbar joint range of motion examination | 2nd week, 4th week, 8th week examination change
  Lumbar joint range of motion examination( flexion-extansion-lateral flexion-rotation)
Physical examination-straight leg raise test | 2nd week, 4th week, 8th week examination change
  straight leg raise test- It is recorded whether there is normal or abnormal
Physical examination-femoral nerve stretch test | 2nd week, 4th week, 8th week examination change
  femoral nerve stretch test - It is recorded whether there is normal or abnormal
Physical examination-Walleix palpation | 2nd week, 4th week, 8th week examination change
  Walleix palpation- It is recorded whether there is tenderness in Walleix palpation.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)